CLINICAL TRIAL: NCT04997018
Title: A Phase II Study of Radiotherapy to the Prostate and Dose Intensification to the Dominant Intra- Prostatic Lesion (DIL) Using Ultra-Hypofractionated, MR-Guided Radiotherapy
Brief Title: A Study of MRI-guided High-dose Radiation Therapy in Prostate Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-308
Record Dates: First submitted 2021-08-04; First posted 2021-08-09 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: SBRT; stereotactic body radiation therapy; prostate cancer; 21-308; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Prostate cancer patients (Experimental): Intermediate-risk prostate cancer patients will be eligible for this study. Risk groups will be assigned as per NCCN guidelines. Intermediate-risk patients will be defined as:
  * PSA 10-20 ng/ml or
  * Gleason score = 7
  * Clinical stage T2b/T2c
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — Patients enrolled in this study will undergo ultra-hypofractionated radiation utilizing MR guided, daily online adaptive planning. Patients will receive a standard dose of 8 Gy/fraction for five fractions for a total dose of 40 Gy to the prostate with a simultaneously-delivered boost of 9 Gy for five fractions (clinically non-standard dose of 45 Gy total) to a single dominant lesion with a maximum dimension of at least 0.5 cm, as determined on the pretreatment diagnostic T2 MRI imaging. In the setting of two similarly-sized "dominant" lesions, both will be boosted.
  Other Names: SBRT

SUMMARY:
One of the usual approaches to treating intermediate-risk prostate cancer is a type of radiation therapy called SBRT (stereotactic body radiation therapy). SBRT delivers higher than standard doses of radiation over a lower number of treatment sessions. However, there is a 20% chance that intermediate-risk prostate cancer will come back after this treatment. The purpose of this study is to find out whether giving an even higher dose (a "boost" dose) of radiation directly to the main tumor and the standard dose of radiation to the rest of the prostate may cure the cancer or prevent it from coming back for a longer period of time while causing few side effects.

ELIGIBILITY:
Inclusion Criteria:

* Intermediate-risk prostate cancer patients will be eligible for this study. Risk groups will be assigned as per NCCN guidelines. Intermediate-risk patients will be defined as:

  * PSA 10-20 ng/ml or
  * Gleason score = 7 or
  * Clinical stage T2b/T2c or
* Additionally, patients will be required to meet all of the following criteria:

  * Age ≥ 18
  * Karnofsky Performance Status (KPS) ≥ 80 (Appendix 1)
  * Prostate size ≤ 80 cc
  * Presence of a T2-visible prostatic lesion with maximum dimension of ≥ 0.5 cm and no more than one additional disease focus
  * MRI findings: Lesion may contact the capsular edge, possible extracapsular extension (ECE) permitted
  * International Prostate Symptom Score ≤ 15
  * Satisfy all MRI screening criteria and be willing to fill out the standard MRI screening form

Exclusion Criteria:

Patient will be excluded if they meet any one of the following criteria:

* Gleason score >7
* PSA >20
* Prior or concurrent androgen deprivation therapy for prostate cancer MRI findings: suspicious for/probable ECE
* MRI findings: >2 disease foci identifiable
* Evidence of metastatic disease on bone scan or MRI/CT
* MRI ineligibility due to: the presence of a cardiac pacemaker, defibrillator, or other implanted metallic or electronic device which is considered MR unsafe; severe claustrophobia; inability to lie flat for the duration of the study; etc.
* Metallic implant or device in the pelvis that might distort the local magnetic field and compromise quality of mp-MRI
* Lateral pelvic separation greater than 50 cm and/or anterior-posterior separation greater than 35 cm which are incompatible with MRCAT reconstruction
* Contra-indications to receiving gadolinium contrast
* KPS < 80
* Pelvic or prostate MRI or CT (MRI preferred) evidence of radiographic T3, T4, or N1 disease
* Prior history of transurethral resection of the prostate
* Prior history of urethral stricture
* Prior history of pelvic irradiation
* History of inflammatory bowel disease
* Unable to give informed consent
* Unable to complete quality of life questionnaires
* Abnormal complete blood count, including any of the following:

  * Platelet count less than 75,000/ml
  * Hb level less than 10 gm/dl
  * WBC less than 3.5/ml
* Abnormal renal function tests (creatinine > 1.5)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-08-04 (Actual); Primary Completion 2026-08-04 (Estimated); Study Completion 2026-08-04 (Estimated)

PRIMARY OUTCOMES:
Comparison of pretreatment biopsy with post-treatment biopsy | 24 months
  The primary outcome of efficacy will be studied using post -treatment biopsies. To demonstrate efficacy of dose escalation to the DIL, the investigators aim to reduce the positive post-treatment biopsy rates at 24 months for intermediate risk disease from 20% to 10%.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Brennan, MBBCH BAO, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering at Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering at Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering at Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering at Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering at Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org